CLINICAL TRIAL: NCT01450605
Title: Korean Post-marketing Surveillance for Reyataz®
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI424-414
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: HIV-1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients ≥ 13 years of age with HIV-1: Patients ≥ 13 years of age with HIV-1 who are on Reyataz® treatment at the time of enrollment and have never been participated in this study previously or who are initiating Reyataz® treatment for the first time in the real-life conditions in its registered indication(s) as required by KFDA
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — Patients are previously on Reyataz® treatment or initiated Reyataz® for the first time

SUMMARY:
The purpose of this post-marketing surveillance is to investigate and confirm the type and incidence of newly identified adverse events and any other factors affecting safety and efficacy of Reyataz® so that the regulatory authority can manage the marketing approval properly

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 13 years of age with HIV-1 who are on Reyataz® treatment at the time of enrollment and have never been participated in this study previously or who are initiating Reyataz® treatment for the first time in the real-life conditions in its registered indication(s) as required by KFDA

Exclusion Criteria:

* According to Warning/Caution in local label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥ 13 years of age with HIV-1 who are on Reyataz® treatment at the time of enrollment and have never been participated in this study previously or who are initiating Reyataz® treatment for the first time in the real-life conditions in its registered indication(s) as required by KFDA
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2011-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Adverse events occurrence | 30 days after last dose of study drug
  Incidence (per person-time) and confidence interval of overall adverse events and each adverse event will be computed per surveillance period

SECONDARY OUTCOMES:
Human Immunodeficiency Virus (HIV) Ribonucleic acid (RNA) level before and after drug administration | Baseline and 16 weeks after first treatment
CD 4 T-cell count before and after drug administration | Baseline and 16 weeks after first treatment
Overall efficacy evaluation by investigator's discretion | Baseline and 16 weeks after first treatment
  Based on laboratory test results including HIV RNA (viral load) and CD4 T-cell count, clinical findings, subjective findings and objective findings in comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx